CLINICAL TRIAL: NCT04023695
Title: Trigger Finger Corticosteroid Injection With and Without Local Anesthetic; a Randomized, Double Blind Controlled Trial
Brief Title: Trigger Finger Corticosteroid Injection With and Without Local Anesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Brian Drolet, Assistant Professor Department of Plastic Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1064521-12
Record Dates: First submitted 2019-07-01; First posted 2019-07-17 (Actual); Results first posted 2019-10-22 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Adrenal Cortex Hormones; Lidocaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid with lidocaine with epinephrine (Active Comparator): This arm includes an injection mixture of corticosteroid and lidocaine with epinephrine
  Interventions: Drug: Corticosteroid with lidocaine with epinephrine
- Corticosteroid with normal saline (Experimental): This arm includes a mixture of corticosteroid and normal saline. The purpose of normal saline is the keep the volume and concentration similar when compared to the injections containing lidocaine.
  Interventions: Drug: Corticosteroid with normal saline

INTERVENTIONS:
Drug: Corticosteroid with lidocaine with epinephrine — Trigger finger injection
  Arms: Corticosteroid with lidocaine with epinephrine
Drug: Corticosteroid with normal saline — Trigger finger injection
  Arms: Corticosteroid with normal saline

SUMMARY:
Steroid injection is the first line treatment for trigger finger. Steroid injection is sometimes mixed with a local anesthetic.

DETAILED DESCRIPTION:
The treatment of trigger finger involves an injection of corticosteroid. Corticosteroid treats the underlying inflammatory pathology. Some surgeons add lidocaine with epinephrine as a local anesthetic with the injection. Lidocaine with epinephrine is associated with a burning sensation and may be the primary pain associated with the injection. We hypothesize that a corticosteroid injection without lidocaine with epinephrine will be less painful, and equally effective in treating trigger finger

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old with trigger finger

Exclusion Criteria:

* Preference for open trigger finger release
* Not a candidate for corticosteroid injection
* Contraindication to lidocaine with epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Corticosteroid With Lidocaine With Epinephrine | Corticosteroid With Normal Saline
Started | 57 | 53
Completed | 57 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid With Lidocaine With Epinephrine | Corticosteroid With Normal Saline | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Continuous [Mean (Full Range); unit: years] | 62.7 [39 to 84] | 66 [35 to 84] | 64.3 [35 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 55 | 50 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 57 | 53 | 110

OUTCOME MEASURES:

1. Primary Outcome: Pain Outcome: Visual Analog Scale
Description: Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever
Time Frame: Assessed 1 minute after injection (in clinic)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Corticosteroid With Lidocaine With Epinephrine | Corticosteroid With Normal Saline
Number analyzed (Participants) | 57 | 53
score on a scale | 3.5 [0 to 7] | 2 [0 to 8]

2. Primary Outcome: Pain Outcome: Visual Analog Scale
Description: Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever
Time Frame: Assessed after 24 hours after injection (by phone)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Corticosteroid With Lidocaine With Epinephrine | Corticosteroid With Normal Saline
Number analyzed (Participants) | 57 | 53
units on a scale | 1.2 [0 to 3] | 1 [0 to 6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Corticosteroid With Lidocaine With Epinephrine | Corticosteroid With Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04023695/Prot_SAP_000.pdf